CLINICAL TRIAL: NCT02574026
Title: MagnetoEncephaloGraphy Study of Cerebral Activations Induced by Psychomotor Tasks for Target Localisation in View of BCI Clinical Trial
Brief Title: Tapfinger Psychomotor Target
Acronym: TAPFINGER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010-A00421-38
Record Dates: First submitted 2015-10-05; First posted 2015-10-12 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Functional Brain Mapping
Keywords: MEG; EEG; MRI; Brain mapping; functional imaging; brain computer interface

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychomotor tasks (Experimental): 20 healthy subjects and 10 tetraplegic patients will participate to acquisition of MEG, EEG, MRI data during a motor tasks
  Interventions: Behavioral: Psychomotor tasks

INTERVENTIONS:
Behavioral: Psychomotor tasks — the acquisition of data will be performed in one unique session no drug administration no surgery

SUMMARY:
The study aims at mapping the magnetoencephalographic (MEG) activities induced in normal volunteers by tapping the finger .

DETAILED DESCRIPTION:
Normal healthy (20) volunteers and tetraplegic patients(10) will be submitted to the temporo-spatial mapping of their brain activity, both sensory and motor, induced by a simple behavioral task, consisting on tapping with the finger on a detection pad. This will be done in a light and then dark environment, on a rythm spontaneous and then paced by sound bips. Accelerometric recording will provide the three dimensionnal displacements of the finger as well as the time code.

Brain activity is simultaneously recorded using MEG (306 channels) and EEG (64 channels. Data will be processed by an INPLS algorithm to detect the predictors of activity, their location and time-course.

3D mapping data will be matched with the patient's anatomy provided by 1.5T MRI previously performed.

The aim of the study is to prepare the strategy of implantation of multielectrodes ECoG implants to restore motility in tetraplegic patients in a human BCI protocol currently under development.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 18 and 70 years
* Informed consent
* Benefiting from Social Security
* French or english speaking, to understand study procedure
* Tetraplegic patients : traumatic injury of the cervical spine with retained respiratory autonomy and without associated head injury

Exclusion Criteria:

* Contra-indication to MRI
* Claustrophobia
* Mental disorders
* Pregancy
* All categories of protected persons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
MEG records for functional brain mapping | one hour study
  This study is not a therapeutic clinical study. No treatment is being delivered.

SECONDARY OUTCOMES:
MEG measurements during psychomotor tasks | one hour study
  MEG records induced by finger tapping will be performed either randomly or following sound bips pacing.
EEG measurements during psychomotor tasks | one hour study
  EEG records induced by finger tapping will be performed either randomly or following sound bips pacing.

CONTACTS AND LOCATIONS:
Overall Officials: Alim L Benabid, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CLINATEC, Grenoble, France